CLINICAL TRIAL: NCT06434441
Title: Radiographic Assessment of Horizontal Bone Augmentation of Full Atrophic Maxillary Alveolar Ridges Using Calvarial Versus Iliac Crest Bone Blocks:
Brief Title: Bone Augmentation Using Calvarial Versus Iliac Crest Bone Blocks.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Amr Gibaly, Associate Professor of Oral and Maxillofacial Surgery, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Bone Atrophy
Keywords: Bone graft; Iliac crest blocks; Calverial bone blocks; Horizontal bone gain

STUDY DESIGN:
Intervention Model Description: A) The Study group:
  The patients within the study group will receive mono-cortical bone block calvarial grafts
  B) The Control group:
  The patients within the control group will receive mono-cortical bone block iliac crest grafts,
Who Masked: Outcomes Assessor
Masking Description: Masking in not applicable for the patients or the operators
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group: (Active Comparator): The patients will receive calverial grafts, to reconstruct the deficient maxillary ridge
  Interventions: Procedure: Autogenous bone augmentation
- Control group: (Active Comparator): The patients will receive iliac crestgrafts, to reconstruct the deficient maxillary ridge
  Interventions: Procedure: Autogenous bone augmentation

INTERVENTIONS:
Procedure: Autogenous bone augmentation — Maxillary alveolar bone reconstruction

SUMMARY:
This study aims to evaluate and compare the quantity of the radiographic horizontal bone gain of severely deficient complete maxillary ridges reconstructed by bone block harvest from the iliac crest versus the calvarial bones

DETAILED DESCRIPTION:
Although the calvarial bones represent a nearby donor site for maxillary augmentation of matching bone origin, the excessive volume of bone needed to reconstruct a severely deficient arch, the limited cancellous bone volume, and the arciform pattern of the skull cap that yield the curvatures of the harvested cortical blocks incompatible with the topography of the maxillary arch, all represent limitations for the calvarial graft.

The anterior iliac crest is frequently used for free bone grafting by being subcutaneous and generous to afford ample bone blocks of favorable curvatures. However, the minute cortical overlay and its endochondral origin contribute to excessive graft resorption. Pikos et al. demonstrated that a reasonable amount of graft resorption could occur with atraumatic surgical intervention and intimate graft fixation.

This study aims to evaluate and compare the quantity of the radiographic horizontal bone gain of severely deficient complete maxillary ridges reconstructed by bone block harvest from the iliac crest versus the calvarial bones.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the clinical and radiographic interpretation of horizontal maxillary ridge deficiency of less than 5 mm

Exclusion Criteria:

* Any previous maxillary reconstructive or dental implant treatment.
* Any local pathologic lesion or systemic disease that would affect the typical pattern of bone healing.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Horizontal bone gain | 6 months consolidation period
  the study compares the horizontal bone gain of reconstructed maxillary alveolar ridges after being augmented with calverial and iliac crest bone grafts radiographically by millimeters

SECONDARY OUTCOMES:
Immunohistochemical bone formation | 6 months consolidation period
  the study compares the bone area percent of the consolidated calverial and iliac crest bone grafts

CONTACTS AND LOCATIONS:
Locations (1):
- Amr Gibaly, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No